CLINICAL TRIAL: NCT04653727
Title: Effects of Interventions and Lifestyle Modifications in Integrative Medicine and the Course of Infectious Respiratory Diseases Including COVID-19
Brief Title: Effects of Integrative Medicine on Infectious Respiratory Diseases Including COVID-19
Acronym: AtemNHK
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, PI, Charite University, Berlin, Germany
Other Study IDs: AtemNHK
Record Dates: First submitted 2020-11-23; First posted 2020-12-04 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Covid19; Influenza A; Respiratory Disease
MeSH Terms: conditions — COVID-19; Respiration Disorders | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Online survey with 3.000 participants using mobile website technology
  Interventions: Other: Cross-sectional survey

INTERVENTIONS:
Other: Cross-sectional survey — No intervention.

SUMMARY:
The outbreak of the novel coronavirus SARS-CoV-2 caused a health emergency of international proportions when it was declared by the World Health Organization (WHO) in January 2020. Since then, the virus has spread internationally and the WHO has classified the outbreak as a pandemic. In the context of the increasing reporting of this pandemic and the increasing governmental measures to limit or slow down the spread of SARS-CoV-2 by all means, there is so far little scientific evidence for the effects of a healthy lifestyle on the disease. The aim of this study is to compare the potential of different, possibly protective lifestyles using the example of the COVID-19 pandemic. We will conduct an online survey with 3.000 participants using mobile website technology.

ELIGIBILITY:
Inclusion Criteria:

- Present declaration of consent

Exclusion Criteria:

- Lack of consent to participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is advertised via a website, thus all interested people can participate in this survey.
Sampling Method: Probability Sample
Enrollment: 1287 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 infection | Assessed retrospectively (last 6 months) with self-designed question

SECONDARY OUTCOMES:
Influenza virus infection | Assessed retrospectively (last 6 months) with self-designed question
Other respiratory infections | Assessed retrospectively (last 6 months) with self-designed question
Dietary habits | Assessed retrospectively (last 6 months) with self-designed question
Sports activity | Assessed retrospectively (last 6 months) with self-designed question
Time spent in nature | Assessed retrospectively (last 6 months) with self-designed question
Use of hydrotherapy/Kneipp applications | Assessed retrospectively (last 6 months) with self-designed question
Use of anthroposophic medicine | Assessed retrospectively (last 6 months) with self-designed question
Use of digital health services | Assessed retrospectively (last 6 months) with self-designed question
Use of phytotherapy | Assessed retrospectively (last 6 months) with self-designed question
Use of dietary supplements | Assessed retrospectively (last 6 months) with self-designed question
WHO-5 Well-Being Index | Assessed when filling out the questionnaire (Baseline)
  The scale ranges from 0 to 100, where 0 is the lowest level of well-being / lowest quality of life and 100 is the highest level of well-being / highest quality of life.
Numeric analog scale (NAS) stress | Assessed retrospectively (last 6 months) with self-designed question
  The NAS ranges from 0 to 10, where 0 is the lowest level of stress and 10 is the highest level of stress.
Numeric analog scale (NAS) anxiety | Assessed retrospectively (last 6 months) with self-designed question
  The NAS ranges from 0 to 10, where 0 is the lowest level of anxiety and 10 is the highest level of anxiety.
Numeric analog scale (NAS) depression | Assessed retrospectively (last 6 months) with self-designed question
  The NAS ranges from 0 to 10, where 0 is the lowest level of anxiety and 10 is the highest level of anxiety.
Use of relaxation / mind body approaches | Assessed retrospectively (last 6 months) with self-designed question
Alcohol consumption | Assessed retrospectively (last 6 months) with self-designed question
Cigarette consumption | Assessed retrospectively (last 6 months) with self-designed question
Self-efficacy | Assessed when filling out the questionnaire (Baseline)
  The scale ranges from 0 to 100, where 0 is the lowest level of self-efficacy and 100 is the highest level of self-efficacy.
Sick leave | Assessed retrospectively (last 6 months) with self-designed question

OTHER OUTCOMES:
Qualitative interviews | Conducted 1 month after completion of the questionnaire (once)

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeitler M, Erehman A, Koppold DA, Ortiz M, Jerzynski L, Stockigt B, Rotter G, Blakeslee S, Brinkhaus B, Michalsen A, Seifert G, Cramer H, Kandil FI, Kessler CS. Self-care and lifestyle interventions of complementary and integrative medicine during the COVID-19 pandemic-A cross-sectional study. Front Med (Lausanne). 2023 Jan 9;9:1033181. doi: 10.3389/fmed.2022.1033181. eCollection 2022. PMID 36698795